CLINICAL TRIAL: NCT07047183
Title: A Single-Arm, Prospective Clinical Study of Venetoclax Combined With Azacitidine Followed by Bridging Transplantation in Patients With High-Risk Myelodysplastic Neoplasms With Increased Blasts 2 (MDS-IB2)
Brief Title: Clinical Study of Venetoclax Combined With Azacitidine as Bridging Therapy Prior to Hematopoietic Stem Cell Transplantation in Patients With Higher-Risk Myelodysplastic Syndromes
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yehui Tan (Other)
Responsible Party: Sponsor-Investigator, Yehui Tan, Professor, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-HS-061
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Myelodysplastic Neoplasms; Transplantation
MeSH Terms: interventions — venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- venetoclax + Azacitidine (Experimental)
  Interventions: Drug: VEN (Venetoclax)

INTERVENTIONS:
Drug: VEN (Venetoclax) — Enrolled patients will receive: Venetoclax: 100 mg on Day 1, 200 mg on Day 2, and 400 mg on Days 3-14. Azacitidine: 75 mg/m² on Days 1-7. Cycle duration: 28 days Total cycles: 1 to 2 cycles
  Other Names: Azacitidine

SUMMARY:
A Single-Arm, Prospective Clinical Study of Venetoclax Combined with Azacitidine Followed by Bridging Transplantation in Patients with High-Risk Myelodysplastic Neoplasms with Increased Blasts 2 (MDS-IB2)

DETAILED DESCRIPTION:
This is a single-center, single-arm, prospective study investigating pre-transplant bridging therapy in patients aged ≥18 years with higher-risk MDS-IB2. The study plans to enroll 46 eligible patients. Participants will receive Venetoclax combined with Azacitidine, administered in 28-day cycles for 1 to 2 cycles. Treatment response will be assessed according to the IWG 2023 HR-MDS response criteria.Patients achieving modified Composite Complete Remission (mCRc: CR or CR-equivalent + CRL + CRh) after Cycle 1 will proceed directly to transplantation. Patients not achieving mCRc will receive a second cycle of therapy. All patients will undergo allogeneic hematopoietic stem cell transplantation (allo-HSCT) within 3 months after completing Cycle 2, regardless of mCRc status. Patients unable to proceed to transplantation will receive standard institutional care and undergo follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed MDS confirmed by morphological and immunophenotypic analysis of bone marrow；
2. Age ≥18 years, any gender；
3. Bone marrow blasts ≥10%；
4. IPSS-R score >4.5；
5. ECOG performance status 0-2；
6. Scheduled for allogeneic hematopoietic stem cell transplantation (allo-HSCT)；
7. Adequate major organ function：

   * Cardiac: LVEF ≥50%
   * Hepatic: Bilirubin ≤1.5×ULN
   * AST/ALT ≤2.5×ULN
   * Renal: Creatinine clearance ≥60 mL/min；
8. Written informed consent provided by the patient or legally authorized representative.

Exclusion Criteria:

1. Extramedullary disease involvement；
2. Hypersensitivity to any study drugs；
3. Clinically significant hepatic/renal dysfunction exceeding inclusion thresholds；
4. Severe cardiac disease, including congestive heart failure, myocardial infarction, and cardiac insufficiency;
5. Concurrent malignant tumors of other organs, which can be enrolled if previously cured;
6. Active tuberculosis or HIV infection;
7. Concomitant hematologic disorders;
8. Pregnancy or lactation;
9. Inability to comply with protocol requirements;
10. Concurrently participating in other clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
2-Year Relapse-Free Survival(2-RFS) | From date of index treatment to death, disease progression, or end of study, whichever came first, assessed up to 24 months.
  Defined as the time from enrollment in this study to the occurrence of relapse. For patients without relapse, the time is calculated until death from any cause or the time of the last follow-up

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of index treatment to death, disease progression, or end of study, whichever came first, assessed up to 48 months.
  Defined as the time from enrollment in this study to death from any cause. If the exact date of death is unknown, the time of death is defined as the last contact date. If the patient is still alive, the last observed time will be used, and the patient's OS will be considered for analysis.
Cumulative Relapse Rate (CIR) | rom date of index treatment to death, disease progression, or end of study, whichever came first, assessed up to 24 months.
  Defined as the proportion of patients who experience disease relapse from the time of enrollment in this study.
Composite Complete Response Rate（mCRc） | Through study completion, an average of 1 year
  Complete Remission (CR) or CR-equivalent+ CR with partial hematologic recovery (CRL) + CR with limited hematologic recovery (CRh)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China